CLINICAL TRIAL: NCT00601848
Title: A Phase II Study of Pleural Photodynamic Therapy for Patients With Non-small Cell Lung Cancer and Pleural Spread
Brief Title: Photodynamic Therapy in Treating Patients With Resectable Non-Small Cell Lung Cancer That Has Spread to the Pleura
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual and change in standards of care
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 05503; CDR0000583050
Record Dates: First submitted 2008-01-25; First posted 2008-01-28 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; malignant pleural effusion
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant | interventions — Drug Therapy; Dihematoporphyrin Ether; Immunohistochemistry; Spectrum Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Photodynamic Therapy (Experimental): PDT
  Interventions: Drug: chemotherapy; Drug: porfimer sodium; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: spectroscopy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: chemotherapy
Drug: porfimer sodium
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: spectroscopy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug, such as porfimer sodium, that is absorbed by tumor cells. The drug becomes active when it is exposed to light. When the drug is active, tumor cells are killed. Giving photodynamic therapy during surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects and how well photodynamic therapy given during surgery works in treating patients with resectable non-small cell lung cancer that has spread to the pleura.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall survival rate of patients with non-small cell lung cancer (NSCLC) and malignant pleural spread treated with standard front-line chemotherapy followed by surgical resection and intra-operative porfimer sodium (Photofrin®)-mediated photodynamic therapy.
* To determine the feasibility and toxicities of standard front-line chemotherapy followed by surgical resection and intra-operative Photofrin®-mediated photodynamic therapy in these patients.

Secondary

* To determine the progression-free survival and pleural progression-free survival of these patients.
* To determine the absolute Photofrin® levels in tumor and normal tissues resected from these patients using spectrofluorometric methods.
* To determine the tumor to normal tissue ratios of Photofrin® in these patients.
* To measure the optical properties of tumor and normal tissues in situ.
* To compare the Photofrin® concentration of tumor and normal tissues made with the in situ measurements to the measurements made with spectrofluorometric method.

OUTLINE: This is a multicenter study.

Patients receive 2-4 courses of standard front-line chemotherapy prior to surgery (if they have not completed the front-line chemotherapy).

Patients receive porfimer sodium (Photofrin®) IV over 5-15 minutes. Approximately 24 hours after receiving porfimer sodium, patients undergo surgery to remove the primary tumor and the pleural disease to a thickness of 5 mm or less*. Patients then undergo intraoperative photodynamic therapy to the residual disease. Some patients may undergo postoperative radiotherapy to the mediastinum and/or surgical scar if clinically indicated.

NOTE: *If the disease cannot be resected to less than 5 mm, PDT will not be delivered

Tumor and normal tissue samples are obtained from the surgical specimen and examined prior to light delivery at the time of thoracotomy, and after light delivery. Tissue samples are analyzed for porphyrin levels using a spectrofluorometric assay of tissue specimens and an in situ optical method intra-operatively. Samples are also assessed for V-cadherin, markers for oxidative stress, markers associated with photosensitizer uptake, markers for angiogenesis, markers for hypoxia, activation of signaling pathway components (including EGFR, p38 MAPK, Akt, and p42/44 MAPK) via immunohistochemistry.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer (NSCLC)

  * Must have clinical and/or pathological evidence of pleural spread
  * Primary tumor must be resectable as assessed by the attending thoracic surgeon
* Patients who have received or are currently receiving two-to-four courses of standard front-line chemotherapy are eligible

PATIENT CHARACTERISTICS:

* Must be medically fit to tolerate surgery
* No CTCAE v3.0 grade III-IV elevations in liver transaminases
* Bilirubin ≤ 1.5 mg/dL
* No known HIV infection
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior treatment for NSCLC except pleurodesis or standard front-line chemotherapy
* No prior pemetrexed disodium chemotherapy
* No prior mantle radiotherapy
* No concurrent chemotherapy or radiotherapy during the active study treatment period

  * Post-operative radiotherapy will be administered as clinically indicated

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-11; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cengel, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Photodynamic Therapy: PDT
  chemotherapy
  porfimer sodium
  immunohistochemistry staining method
  laboratory biomarker analysis
  spectroscopy
  therapeutic conventional surgery
Period: Overall Study
Arm/Group | Photodynamic Therapy
Started | 9
Completed | 0
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: PDT
  chemotherapy
  porfimer sodium
  immunohistochemistry staining method
  laboratory biomarker analysis
  spectroscopy
  therapeutic conventional surgery
Arm/Group | Single Arm
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Assessment of Pleural Photodynamic Therapy
Description: Toxicities of PDT as defined by CTCAE v4.0
Time Frame: One year
Population: The study was terminated. Despite all possible efforts to contact the PI/study team members, no data are available to be reported
Arm/Group | Single Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Survival
Description: Subject survival post PDT
Time Frame: 5 years
Population: as for outcome 1
Arm/Group | Single Arm
Number analyzed (Participants) | 0

3. Primary Outcome: Pleural Progression-free Survival
Description: Amount of time from PDT to disease progression in pleura
Time Frame: 5 years
Population: as for outcome 1
Arm/Group | Single Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: Amount of time from PDT to disease progression at any site in the body
Time Frame: 5 years
Population: as for outcome 1
Arm/Group | Single Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: Photofrin® Uptake
Description: Measured uptake of PDT drug
Time Frame: 90 days
Population: as for outcome 1
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes